CLINICAL TRIAL: NCT04049734
Title: Evaluation of Oral Losartan in the Prevention of Post-ERCP Pancreatitis
Brief Title: Oral Losartan in Prevention of Post-ERCP Paancreatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shereen Abou Bakr Saleh, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 689
Record Dates: First submitted 2019-08-03; First posted 2019-08-08 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Post-ERCP Acute Pancreatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients received the oral losartan (Active Comparator): 50 patients with obstructive jaundice indicated for ERCP and received oral losartan 1 hour before ERCP as a prophylaxis of post-ERCP pancreatitis
  Interventions: Drug: oral losatan
- patients didn't receive the oral losartan (No Intervention): 50 patients with obstructive jaundice indicated for ERCP and didn't receive any prophylactic drugs

INTERVENTIONS:
Drug: oral losatan — 50 mg of oral losartan one hour before the ERCP once
  Arms: patients received the oral losartan

SUMMARY:
Oral losartan given in the dose of 50 mg one hour before ERCP was studied in the prevention of post ERCP pancreatitis in 50 patients indicated for ERCP in comparison with another 50 patients underwent ERCP without receiving oral losartan.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient indicated for ERCP
* Patients with obstructive jaundice.
* Patients with dilated intra-hepatic or extra-hepatic bile ducts due to malignant or benign lesions.

Exclusion Criteria:

* Patients refusing to undergo the procedure or signing the informed consent
* Patients with clinically evident acute pancreatitis before the procedure
* Patients with previous endoscopic or surgical sphincterotomy
* Patients with current use of losartan
* Patients who are allergic or hypersensitive to losartan or hydro soluble contrast solutions
* Patients receiving NSAIDS within a week prior to assessment
* Patients with severe co-morbid conditions as cardiovascular disease, renal failure or decompensated liver cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with development of acute pancreatitis | 24 hours
  Number of participants with development of abdominal pain and elevated serum amylase and/or lipase